CLINICAL TRIAL: NCT02787148
Title: The Impact of Psychotherapy on Hemodynamic and Inflammatory Risk Factors for Cardiovascular Disease in Major Depression
Brief Title: Psychotherapy and Cardiovascular Risk Factors in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Dr. rer. nat. Frank Euteneuer, PhD, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFG EU 154 2 1
Record Dates: First submitted 2016-02-10; First posted 2016-06-01 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Depression
Keywords: cognitive behavioral therapy; psychotherapy; cardiovascular health; psychoneuroimmunology
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral therapy (Experimental): Cognitive behavioral therapy for Major Depression
  Interventions: Behavioral: Cognitive behavioral therapy
- Waitlist group (No Intervention): Waitlist group to control for repeated physiological measures and fluctuations over time

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy
  Arms: Cognitive behavioral therapy

SUMMARY:
Prospective studies indicate that patients with depression are at increased risk for cardiovascular disease. Depression is also associated with a number of hemodynamic features, which are known risk factors for cardiovascular morbidity such as increased heart rate, reduced heart rate variability and blood pressure alterations. These hemodynamic alterations may explain in part the increased cardiovascular risk associated with depression.

The purpose of this study is to determine whether treatment for depression with cognitive behavior therapy (CBT) is effective in reducing hemodynamic cardiovascular risk factors. Hemodynamic assessments including heart rate, heart rate variability, continues blood pressure, blood pressure variability, baroreceptor sensitivity and peripheral vascular resistance will be conducted at baseline, after treatment and 2-month follow up. In addition, circadian hemodynamic variations such as 24-hour heart rate variability, nocturnal blood pressure dipping and immunological biomarkers will be assessed. Eighty patients with Major Depression will be randomly assigned to either a CBT treatment condition (14 hour-long, weekly sessions) or a waitlist condition, to control for potential changes in hemodynamic parameters without any intervention and the impact of repeated-measurement.

ELIGIBILITY:
Inclusion Criteria:

* patients with Major Depression (DSM IV), BDI >=14
* age:18-65 years
* patients without antidepressive medication (stable for at least 2 weeks)
* comorbidity with other psychiatric disorders is permitted, as far as depressive symptoms are dominating

Exclusion Criteria:

* current psychotherapy
* psychotic disorder
* serious drug-addiction
* drugs which seriously affect immune status (except contraceptives) or central
* nervous system functions (except antidepressants)
* infections during the last 2 weeks
* injuries during the last 2 weeks
* neurological disorders
* diseases which affect immune status or central nervous system functions (e.g. rheumatoid arthritis, CVD,etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms (BDI-II) | Change from baseline (beginning of therapy) to 3 month after baseline, to 2-month-follow up

SECONDARY OUTCOMES:
Change in heart rate variability | Change from baseline (beginning of therapy) to 3 month after baseline, to 2-month-follow up
Change in blood pressure | Change from baseline (beginning of therapy) to 3 month after baseline, to 2-month-follow up
Change in baroreceptor sensitivity (ms/mmHg) | Change from baseline (beginning of therapy) to 3 month after baseline, to 2-month-follow up
Change in peripheral vascular resistance (dyne*s/cm5) | Change from baseline (beginning of therapy) to 3 month after baseline, to 2-month-follow up
Change in C-reactive protein | Change from baseline (beginning of therapy) to 3 month after baseline, to 2-month-follow up
Change in proinflammatory cytokines | Change from baseline (beginning of therapy) to 3 month after baseline, to 2-month-follow up
Change in anti-inflammatory interleukin-10 | Change from baseline (beginning of therapy) to 3 month after baseline, to 2-month-follow up
Change in Subjective social status (MacArthur scale) | Change from baseline (beginning of therapy) to 3 month after baseline, to 2-month-follow up

CONTACTS AND LOCATIONS:
Overall Officials: Frank Euteneuer, PhD, Principal Investigator — Department of Clinical Psychology and Psychothearpy, Philipps University of Marburg
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Philipps University Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No